CLINICAL TRIAL: NCT03133143
Title: The Impact of Video Gaming on Cognitive Functioning in People With Schizophrenia
Brief Title: Video Games Among People With Schizophrenia
Acronym: GAME-S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: University of Helsinki (Other); University of Turku (Other); Kowloon Hospital, Hong Kong (Other); Pamela Youde Nethersole Eastern Hospital (Other); Maxgrace Fuller House (Unknown); The Mental Health Association of Hong Kong (Other); Sichuan University (Other)
Responsible Party: Principal Investigator, Maritta Anneli Välimäki, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HSEARS20161228002
Record Dates: First submitted 2017-04-18; First posted 2017-04-28 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Cognitive Function; Schizophrenia and Disorders With Psychotic Features
Keywords: Cognitive Function; Schizophrenia and Disorders with Psychotic Features; Computers, Digital
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: A controlled, single-blind clinical trial with a pragmatic, three-arm parallel-group design.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The sequences of allocation will be concealed until interventions will be assigned. Allocation will not be masked to the researchers, who will recruit patients. Outcome assessors (who will not participate in patient randomisation or daily clinical treatment at the same unit) will be masked. The data analyst (the trial statistician) will be kept blinded to the allocation. Allocation: Randomized The trial manager will allocate the patient to one of the three arms of the trial based on a list of computer-generated random numbers (provided by an external clinical trial randomisation service).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognifit (Experimental): Participants are instructed to play CogniFit 45-60 minutes, 5 days/week. A minimum of 50 gaming hours will be acquired to ensure observable neuroplasticity in the brain after gaming.
  Interventions: Behavioral: Cognifit
- SIMS 4 (Maxis, Inc) (Active Comparator): Participants are instructed to play SIMS 4 45-60 minutes, 5 days/week. A minimum of 50 gaming hours will be acquired to ensure observable neuroplasticity in the brain after gaming.
  Interventions: Behavioral: SIMS 4 (Maxis, Inc)
- Treatment as usual (No Intervention): No specific intervention will be offered to those who receive treatment as usual according to their treatment schedule. The participants are encouraged not to play video games during the study period.

INTERVENTIONS:
Behavioral: Cognifit — CogniFit is an Internet browser-based digital brain training program, to improve cognitive abilities based on a personalised brain training regimen. Participants are instructed to play all games assigned by cognifit from three categories (memory, spatial perception, and mental planning) during each training session. After playing the games in these three categories, they are free to choose which exercises they wish to play.
  Arms: Cognifit
Behavioral: SIMS 4 (Maxis, Inc) — The Sims 4 is a life simulation PC game. It is purely an entertainment game without known cognitive or health-related outcomes. Does not iclude high-intensity action and competition. This specific game and non-competitive games like it in general do not improve attention, working memory, or other cognitive abilities despite being engaging and fun.
  Arms: SIMS 4 (Maxis, Inc)

SUMMARY:
The investigators aim to establish a research project to test the impact of gaming by carrying out a digital gaming interventions, monitoring its cognitive and clinical outcomes, while concurrently performing a multimodal brain imaging experiment.

DETAILED DESCRIPTION:
The effectiveness of the gaming intervention will be assessed using a controlled, controlled, single-blind clinical trial with a pragmatic, three-arm parallel-group design.

Interventions: Participants will be randomised into three groups: Cognitive training (intervention group, CogniFit, N=78), entertainment video gaming (active control group, SIMS4, N=78) and treatment as usual (a passive control group, N=78). The mechanism of CogniFit (intervention) lies on the evidence for computerised exercises focusing on auditory and verbal processing, which are likely to yield improved verbal learning and memory and activate reward systems of the brain that drive brain plasticity in adults with schizophrenia. SIMS4 game (active control) offers entertainment without any known cognitive or health-related outcome. The data collection, subject recruitment and training will be carried out in an outpatient psychiatric units or outpatient clinics, mental health associations, and residential homes in Hong Kong. The study is aimed for patients' diagnoses of schizophrenia.

Recruitment: An extended informed consent process will be used. The health service's medical records at the study site will be screened by the authority of the staff of the organisation. Patients will be screened to determine their eligibility for study participation. Eligible participant will first receive a short leaflet of the study from the staff or during a short information session organised for the participants to consider their availability. If an eligible patient shows interest, more detailed written and oral information will be shared.

After signing informed consent forms (two identical copies), baseline data with background information, Intelligence Quotient (IQ, if available) and MMSE will be collected to show evidence of the participants' capacity to give informed consent. Medication dosage [chlorpromazine equivalence] will be collected as some medications currently used in schizophrenia may affect the response to cognitive training strategies.

Recruitment will continue until the required sample size has been obtained.

Randomisation: After baseline data collection, the Trial Manager will be informed (by email, text message, WhatsApp) about a new participant and he/she will allocate the participant to one of the three arms based on a list of computer-generated random numbers provided by an external clinical trial randomisation service (blocks of 6 consecutive patients, a 1:1:1 ratio). Allocation will be masked to the outcome assessors, and the trial statistician, but it cannot be masked from the RAs who recruit the patients and the treatment staff working with the patients.

For neuroimaging assessment (EEG, fMRI, resting state), a sub-sample from our total sample will be randomised at baseline. Randomisation will be based on a list of computer-generated random numbers.

Power analysis and sample size: The investigators calculated the sample size based on (1) the number of actual pairwise tests to be made for the efficacy of the primary outcome and (2) the two-level modelling approach in the final data analysis, in which the type I error has been adjusted. The statistical efficiency will be ensured using the MANOVA method for multiple group comparison. First, given that video gaming is a fairly novel strategy, the investigators will base the sample size calculation (a priori) on a cognitive-efficacy meta-analysis for patients with schizophrenia showing and overall effect size (ES, Cohens' D) of 0.58 on verbal working memory (a primary outcome). Based on our hypothesis, the primary endpoints are the effects in verbal working memory at 3 and 6 months of cognitive training in the gaming group, in comparison with the other two groups: cognitive training vs. entertainment gaming, cognitive training vs. non-gaming control group. Four pairwise interactions between the contrast of the two comparisons and the two time points will be tested. For multiple comparison tests of four, for a type I error level of 5% (two-sided), an adjusted significant level should be = (1- (1- 0.05)4) /2 = 0.01274 /2 = 0.0064, and the corresponding z score for a one-sided test is 2.49. Given the effect size 0.58, assuming equal sample size of the three groups, with a statistical power of 0.8 and = 0.01274, the investigators require at least 198 subjects (66 per group) by applying the equation, 2(Z1- + Z1- /2)2 / ES2. According to a meta-analysis,40 the total sample size in previous cognitive training studies has typically been 50 (range 10-138).

Using evidence-based rationale for patient flow in this study, the investigators can assume that about 60% of patients that will be screened will not be eligible for the study due to age or lack of capacity to participate in the study. Based on the literature, about 45% of patients with schizophrenia will refuse to participate in the RCT studies, and 16% will drop-out during the course of intervention. Thus, the investigators need a total of 234 participants to be randomply allocated to three study groups, and 198 participants in follow-ups. Based on this knowledge, a total of 985 subjects need to be approached. The numbers are realistic given that the total number of patients with schizophrenia in our study sites is about 5,500, and the total number of schizophrenia patients in Hong Kong is 40,000.

Second, for neuroimaging assessment, a sub-sample of 126 participants from our total sample (N = 198) will need (63%) to be randomised at baseline. Randomisation will be based on a list of computer-generated random numbers. The investigators assume that 30% will drop-out between baseline and the 3-month follow-up assessment, which leave us with 29 patients in each group (totally 87 participants at baseline). The sample size will be appropriate for our neuroimaging assessment; the average number of participants in RCT studies assessing patient cognition or changes in brain structure has been about 20.

The investigators will also verify whether the interventions have been delivered as designed (intervention fidelity). Therefore, patient gaming logs (gaming frequency [number of gaming sessions per week], the length of each session [minutes], number of drop-outs) and patient gaming diaries including descriptions of possible strengths and limitations of the interventions will be analysed with the content analysis based on the data to be collected from patient diaries.

ELIGIBILITY:
Inclusion criteria:

* patients' diagnoses of schizophrenia (Diagnostic and Statistical Manual DSM-IV)
* able to speak Cantonese
* be unfamiliar with video games or at least non-active game players (play < 5h/week)
* have the ability to provide written informed consent
* be viewed as being able to safely take part and have the cognitive status deemed suitable for participation (assessed by a chief psychiatrist based on his/her clinical expertise)

Exclusion criteria:

* meeting diagnostic criteria for a current major depressive, manic or hypomanic episode (DSM-IV), or mental retardation
* having severe visual impairment
* being an active game player (i.e. gaming > 5 h/week)
* displaying a lack of ability to decide their own participation
* displaying substance abuse (other than nicotine dependence)
* having head injury, hemiplegia, or other neurological disorders
* having had an Electroconvulsive Therapy (ECT) in the past six months
* having a lack of Magnetic Resonance Imaging (MRI) compatibility (for example, patients with cardiac pacemakers, metallic implants, restless behaviour)
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Verbal working memory function at 3-month and 6-month follow-ups | 3-month and 6-month follow-ups
  Measured by Letter-number-span task from Wechsler Memory Scale III (WMS III), simplified/traditional Chinese versions. The instrument includes the National Institute of Mental Health - Measurement and Treatment Research to Improve Cognition in Schizophrenia 50 battery (NIMH-MATRICS50).

SECONDARY OUTCOMES:
Cognitive functioning: speed of processing | Baseline, after intervention (three months) and at six months follow-up
  A battery of cognitive tests: speed of processing [Trail Making Test A].
Cognitive functioning: attention | Baseline, after intervention (three months) and at six months follow-up
  A battery of cognitive tests: attention (serotonin transporter; SERT).
Cognitive functioning: vigilance | Baseline, after intervention (three months) and at six months follow-up
  A battery of cognitive tests: vigilance [SERT].
Cognitive functioning: visuo-spatial working memory | Baseline, after intervention (three months) and at six months follow-up
  A battery of cognitive tests: visuo-spatial working memory [Spatial span from WMS III].
Cognitive functioning: reasoning | Baseline, after intervention (three months) and at six months follow-up
  A battery of cognitive tests: reasoning [Wisconsin Card Sorting Task).
Cognitive functioning: problem solving | Baseline, after intervention (three months) and at six months follow-up
  A battery of cognitive tests: problem solving [Wisconsin Card Sorting Task).
Social functioning: severity of social phobia | Baseline, after intervention (three months) and at six months follow-up
  A Chinese version of Brief Social Phobia Scale (BSPS51) assessing severity of social phobia.
Social functioning: treatment response in social phobia | Baseline, after intervention (three months) and at six months follow-up
  A Chinese version of Brief Social Phobia Scale (BSPS51) assessing treatment response in social phobia.
Experience of pleasure: anticipatory component | Baseline, after intervention (three months) and at six months follow-up
  The 'temporal Experience of Pleasure Scale' (TEPS, Chinese version) covers the anticipatory component.
Experience of pleasure: consummatory component | Baseline, after intervention (three months) and at six months follow-up
  The 'temporal Experience of Pleasure Scale' (TEPS, Chinese version) covers the consummatory component.
Self-efficacy | Baseline, after intervention (three months) and at six months follow-up
  Chinese version of 'General Self-Efficacy Scale' (GSE) is a self-report measure of self-efficacy.
Psychotic symptoms | Baseline, after intervention (three months) and at six months follow-up
  The Chinese version of the Clinical Assessment Interview for Negative Symptoms (CAINS) administered by qualified psychiatrists in Hong Kong who have received proper training for this assessment tool.
Anhedonia symptoms | Baseline, after intervention (three months) and at six months follow-up
  Other symptoms, which might confound negative symptom presentation and need to be assessed include: 'The Calgary Depression Scale for Schizophrenia' (CDS-C), an observer-rated Likert-scale to measure depressive symptoms; The Simpson-Angus Rating Scale (SAS), the Barnes Akathisia Rating Scale (BARS), and the Abnormal Movement Involuntary Scale (AIMS).
Avolition symptoms | Baseline, after intervention (three months) and at six months follow-up
  Other symptoms, which might confound negative symptom presentation and need to be assessed include: 'The Calgary Depression Scale for Schizophrenia' (CDS-C), an observer-rated Likert-scale to measure depressive symptoms; The Simpson-Angus Rating Scale (SAS), the Barnes Akathisia Rating Scale (BARS), and the Abnormal Movement Involuntary Scale (AIMS).
Neurocognition: the impact of gaming on brain functional networks (EEG/rsfMRI) | Baseline, after intervention (three months)
  EEG/Resting states fMRI. The impact of gaming on brain functional networks can be revealed by recording neuronal activity with M/EEG during the execution of a working memory task and also during resting-state conditions, which reveal changes in spontaneous activities in the brain.
Neurocognition: the impact of gaming on changes in neuronal dynamics (EEG/rsfMRI) | Baseline, after intervention (three months)
  EEG/Resting states fMRI. The impact of gaming on changes in neuronal dynamics can be revealed by recording neuronal activity with M/EEG during the execution of a working memory task and also during resting-state conditions, which reveal changes in spontaneous activities in the brain.
Neurocognition: the impact of gaming on brain functional networks (EEG/Structural magnetic resonance imaging) | Baseline, after intervention (three months)
  Structural magnetic resonance imaging. The impact of gaming on brain functional networks can be revealed by recording neuronal activity with M/EEG during the execution of a working memory task and also during resting-state conditions, which reveal changes in spontaneous activities in the brain.
Neurocognition: the impact of gaming on changes in neuronal dynamics (EEG/Structural magnetic resonance imaging) | Baseline, after intervention (three months)
  Structural magnetic resonance imaging. The impact of gaming on changes in neuronal dynamics can be revealed by recording neuronal activity with M/EEG during the execution of a working memory task and also during resting-state conditions, which reveal changes in spontaneous activities in the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Maritta Välimäki, Professor, Principal Investigator — Xiang Nursing School, Central South University; Hong Kong Polytechnic University; University of Turku
Locations (9):
- Hong Kong (9):
  - Comfort Rehabilitation Home, Hong Kong
  - Everbright Rehabilitation Centre, Hong Kong
  - Home of Treasure, Hong Kong
  - Kowloon Hospital, Hong Kong
  - Mental Health Association of Hong Kong, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Parklane Rehabilitation Home, Hong Kong
  - Richmond Fellowship of Hong Kong, Hong Kong
  - Maxgrace Fuller House, Kowloon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valimaki M, Yang M, Lam YTJ, Lantta T, Palva M, Palva S, Yee B, Yip SH, Yu KD, Chang HCC, Cheng PYI, Bressington D. The impact of video gaming on cognitive functioning of people with schizophrenia (GAME-S): study protocol of a randomised controlled trial. BMC Psychiatry. 2021 Jan 18;21(1):46. doi: 10.1186/s12888-020-03031-y. PMID 33461506